CLINICAL TRIAL: NCT00168077
Title: Efficacy and Tolerance of BERIPLEX® P/N in Subjects With Acquired Deficiency of Coagulation Factors II, VII, IX and X Due to Oral Anticoagulation
Brief Title: Prothrombin Complex Concentrate for Anticoagulant Reversal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Global Head Clinical Research & Development, CSL Behring
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE1116_3001
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Acquired Coagulation Factor Deficiency
Keywords: Prothrombin Complex Concentrate; Anticoagulant reversal
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

INTERVENTIONS:
Drug: Prothrombin Complex Concentrate

SUMMARY:
Patients on oral anticoagulants need rapid reversal of the anticoagulant effect in case of acute bleeding or emergency surgery. Prothrombin Complex Concentrates are known to provide a fast reversal of the anticoagulant effect, with several advantages over alternatives like vitamin K or FFP.The planned clinical Phase III study is designed to provide clinically relevant data on efficacy and safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects on oral anticoagulation requiring rapid reversal due to acute bleeding or emergency surgery
* INR > 2 at baseline

Key Exclusion Criteria:

* Acute thromboembolic event
* Treatment with any other investigational drug in the last 30 days before study entry
* Less than 2 weeks of stable oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Rapid reversal of anticoagulatory effect

SECONDARY OUTCOMES:
Clinical efficacy assessment (hemostatic effect)
Increase of coagulation factors

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Pabinger-Fasching, Prof., Principal Investigator — Universitätsklinik für Innere Medizin I der Stadt Wien
Locations (15):
- Austria (2):
  - Clinical Trials Registration Coordinator, Feldkirch
  - Clinical Trials Registration Coordinator, Vienna
- Germany (5):
  - Clinical Trials Registration Coordinator, Halle
  - Clinical Trials Registration Coordinator, Hanover
  - Clinical Trials Registration Coordinator, Leipzig
  - For information on sites in Europe, please contact our clinical research team in, Marburg
  - Clinical Trials Registration Coordinator, München
- Hungary (2):
  - Clinical Trials Registration Coordinator, Győr
  - Clinical Trials Registration Coordinator, Veszprém
- Clinical Trials Registration Coordinator, Haifa, Israel
- Lithuania (2):
  - Clinical Trials Registration Coordinator, Kaunas
  - Clinical Trials Registration Coordinator, Vilnius
- Clinical Trials Registration Coordinator, Amsterdam, Netherlands
- Clinical Trials Registration Coordinator, Warsaw, Poland
- Clinical Trials Registration Coordinator, Zurich, Switzerland

REFERENCES:
- [Result] Pabinger I, Brenner B, Kalina U, Knaub S, Nagy A, Ostermann H; Beriplex P/N Anticoagulation Reversal Study Group. Prothrombin complex concentrate (Beriplex P/N) for emergency anticoagulation reversal: a prospective multinational clinical trial. J Thromb Haemost. 2008 Apr;6(4):622-31. doi: 10.1111/j.1538-7836.2008.02904.x. Epub 2008 Jan 15. PMID 18208533
- [Result] Pabinger I, Tiede A, Kalina U, Knaub S, Germann R, Ostermann H; Beriplex P/N Anticoagulation Reversal Study Group. Impact of infusion speed on the safety and effectiveness of prothrombin complex concentrate: a prospective clinical trial of emergency anticoagulation reversal. Ann Hematol. 2010 Mar;89(3):309-16. doi: 10.1007/s00277-009-0830-7. Epub 2009 Sep 29. PMID 19787352